CLINICAL TRIAL: NCT06942559
Title: Brain-Oscillation Synchronized Stimulation of the DMPFC: A Single-Blind Study for Personalized Neuromodulation in OCD
Brief Title: Brain-Oscillation Synchronized Stimulation of the DMPFC
Acronym: BOSS-OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Brigitte Zrenner, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104-2023
Record Dates: First submitted 2025-02-21; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Obsessive Compulsive Disorder (OCD); Treatment Resistant Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Treatment Resistant Obsessive Compulsive Disorder; Transcranial Magnetic Stimulation; Repetitive Transcranial Magnetic Stimulation; Electroencephalography; Electroencephalography Triggered rTMS; EEG-Triggered rTMS; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The clinical trial uses a prospective, randomized, single-blind, two-arm interventional controlled study design to evaluate two treatment arms at a single study site. We aim to recruit 48 adults with a primary diagnosis of Obsessive Compulsive Disorder (OCD).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized, EEG-triggered rTMS (Experimental)
  Interventions: Device: EEG-Triggered Repetitive Transcranial Magnetic Stimulation (rTMS)
- Non-personalized, non-EEG triggered rTMS (Active Comparator)
  Interventions: Device: Non-EEG Triggered Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: EEG-Triggered Repetitive Transcranial Magnetic Stimulation (rTMS) — The rTMS intervention will be delivered using the MagPro XP - Orange Edition stimulator and COOL D-B80 coil to the dorsomedial prefrontal cortex 4 cm anterior to the foot hotspot. EEG data will be analyzed in real-time using the bossdevice MEDICAL and TMS pulses will be synchronized to the negative peak of the frontoparietal theta oscillation.
  500 consecutive EEG theta-oscillation negative-peak triggered quadruplet bursts with a 5 ms inter-pulse interval will be applied at an average inter-burst interval of 2 s. The therapeutic intervention consists of 30 sessions of 2000 TMS pulses each for a total duration per treatment session of 17 minutes.
  Other Names: Personalized rTMS; EEG-triggered rTMS; Personalized TMS; EEG-triggered TMS
  Arms: Personalized, EEG-triggered rTMS
Device: Non-EEG Triggered Repetitive Transcranial Magnetic Stimulation (rTMS) — The rTMS intervention will be delivered using the MagPro XP - Orange Edition stimulator and COOL D-B80 coil to the dorsomedial prefrontal cortex 4 cm anterior to the foot hotspot.
  High-frequency rTMS consisting of 50 trains at 20 Hz (2 s on, 18 s off) will be delivered. The therapeutic intervention consists of 30 sessions of 2000 TMS pulses each for a total duration per treatment session of 17 minutes.
  Other Names: Standard rTMS; Standard TMS; rTMS; TMS
  Arms: Non-personalized, non-EEG triggered rTMS

SUMMARY:
This trial aims to obtain initial evidence about the clinical efficacy and modulation of neurophysiological markers in obsessive compulsive disorder (OCD) using personalized (i.e., electroencephalography (EEG)-triggered) repetitive transcranial magnetic stimulation (rTMS) as compared to non-personalized (i.e., non-EEG triggered), standard rTMS applied to the dorsomedial prefrontal cortex.

DETAILED DESCRIPTION:
This trial uses a prospective, randomized, single-blind study design with two treatment arms at the Centre for Addiction and Mental Health (CAMH) in Toronto, ON. The study aims to compare the clinical effects of EEG-triggered, personalized rTMS (i.e., experimental arm) in the treatment of OCD to those of non-EEG triggered, non-personalized rTMS (i.e., active-comparator arm). Additionally, the study aims to compare the modulation of neurophysiological (i.e., EEG) markers of OCD between the two arms.

Study treatment will be administered five days per week across a six-week treatment course for a total of 30 sessions. Both rTMS arms will use the same TMS coil, stimulation intensity, number of pulses, and anatomical target (i.e., dorsomedial prefrontal cortex).

Clinical outcomes will be measured using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) with clinical response defined as a ≥30% improvement on the Y-BOCS. The self-reported revised Obsessive Compulsive Inventory (OCI-R) and Clinical Global Impressions - Improvement (CGI-I) scale will also be used. Neurophysiological outcomes will be measured by the change in frontoparietal theta amplitude (i.e., 4-7 Hz) and power of TMS-induced theta oscillations.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18-65 years old;
2. Have OCD as a primary disorder, confirmed by a Mini-International Neuropsychiatric Interview (MINI) diagnosis of OCD, with treatment resistance defined as a failure of at least one course of cognitive-behavioural therapy or a single trial of an SSRI;
3. Does not meet criteria for substance use disorder as determined by the MINI (with the exception of nicotine and caffeine);
4. Have a Y-BOCS score >20;
5. Are fluent in the English language (spoken, written, reading);
6. Have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening;
7. Must be deemed to have capacity to provide informed consent;
8. Must sign and date the informed consent form;
9. Stated willingness to comply with all study procedures.

Exclusion Criteria:

1. Have any contraindications to TMS as determined by the Transcranial Magnetic Stimulation Adult Safety Screen (TASS) questionnaire;
2. Have a history of a medical or neurological disorder that affects the central nervous system (e.g., traumatic brain injury, stroke, Parkinson's disease);
3. Are pregnant or breast feeding. TMS is not unsafe in pregnancy and therefore the study team is not requiring a pregnancy test prior to entry. If participants become pregnant during the study they will not be excluded. The study team is not including people who are currently aware of being pregnant as OCD can be affected during the later stages of pregnancy and therefore is a potential confound;
4. Have a history of seizures;
5. Have any metal implants or dentures;
6. Have a serious or unstable medical condition requiring immediate investigation or treatment (e.g., severe or recent cardiac disease);
7. Have a cardiac pacemaker, cochlear implants, implanted electronic devices, non-electronic metallic implants, or other contraindications for rTMS;
8. Take more than 2mg of lorazepam or equivalent benzodiazepine, or any anticonvulsant medication;
9. Fulfill criteria for Alcohol Use Disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | From screening to the end of the follow-up period (1 week post-intervention)
  The Y-BOCS is used to (a) qualify OCD symptoms using a symptom checklist and (b) assess their severity using a symptom severity rating scale. The checklist allows the participant to identify the thoughts and behaviours that are part of their OCD. The severity scale assesses five dimensions of obsessions and compulsions: time spent or occupied, interference with functioning or relationships, degree of distress, resistance, and control (i.e., success with resistance). The scale ranges from 0-40; a lower score indicates less severe OCD, while a higher score indicates more severe OCD.

SECONDARY OUTCOMES:
Obsessive Compulsive Inventory - Revised (OCI-R) | From screening to the end of the follow-up period (1 week post-intervention)
  The OCI-R is a self-reported 18-item scale that measures symptom severity across six domains of OCD: washing, checking, ordering, neutralizing, obsessing, and hoarding. The scale ranges from 0-72; lower scores indicate less severe OCD (or a subclinical presentation for scores <21), while higher scores indicate more severe OCD.
Clinical Global Impressions - Improvement (CGI-I) Scale | From screening to the end of the follow-up period (1 week post-intervention)
  The CGI-I is a clinician-determined assessment that rates change in global clinical presentation (i.e., improvement or worsening) from the baseline presentation on a 7-point scale.
Electroencephalography (EEG) Markers of OCD | From screening to the end of the follow-up period (1 week post-intervention)
  1. Amplitude of frontoparietal theta oscillations in the resting EEG before and after single treatment sessions measured in dB
  2. the power of TMS-induced oscillations in the theta range throughout the six-week treatment course measured in dB

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Zrenner, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this project may be used for future research by internal and/or external project collaborators upon participant consent.
Supporting Information: Study Protocol, SAP